CLINICAL TRIAL: NCT06231420
Title: Daily Step Count Using Pedometer for Sarcopenic Management in Patient With Cirrhosis: Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si 085/2023
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Sarcopenia; Cirrhosis, Liver; Daily Step Count
Keywords: Sarcopenia; Liver cirrhosis; Daily step count; Pedometer recording
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encourage using pedometer group. (Active Comparator): Sarcopenic cirrhotic patient who received pedometer recording and was encouraged to use actively.
  Interventions: Other: Encourage using pedometer; Device: pedometer
- Discourage using pedometer group. (Placebo Comparator): Sarcopenic cirrhotic patient who received pedometer recording but without encouraged to use.
  Interventions: Device: pedometer

INTERVENTIONS:
Other: Encourage using pedometer — Sarcopenic cirrhotic patient used pedometer recording actively with encourage by care provider or investigator
  Arms: Encourage using pedometer group.
Device: pedometer — pedometer

SUMMARY:
The goal of clinical trial is to compare using pedometer in sarcopenic cirrhotic patients. The main questions it aims to answer are:

1. Did the encourage using pedometer group had higher change of skeletal muscle index (SMI) than discourage using pedometer group?
2. How many of patients who had sarcopenic improvement in both groups at 6 months after enrollment?
3. What is the mortality rate and hospital admission in both groups at 12 months after enrollment?

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 - 75 years old
* 2. Cirrhotic patient with diagnosed sarcopenia
* 3. Patients or caregiver who can write and announce Thai language
* 4. Cirrhotic patient who was post liver transplantation > 1 year

Exclusion Criteria:

* 1. Cirrhosis Child-Turcotte-Pugh (CTP) C > 10 2. Refractory ascites 3. Decompensated comorbidity: heart failure NYHA III-IV, ESRD with dialysis, COPD Gold D 4. Performance status ECOG 3-4 5. Bone fracture within 4 weeks or limitation of activity 6. Pregnancy and breastfeeding 7. HCC during treatment with TACE or microwave ablation or radiofrequency ablation within 6 months before enrollment 8. Advanced stage malignancy 9. Received chemotherapy 10. Muscle weakness disease 11. Recent cerebrovascular disease within 6 months and motor weakness grade < II 12. Age 65-75 years old with history of falling > 2 times/year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To compare change of skeletal muscle index (SMI) between encourage using pedometer group and discourage using pedometer group. | 6 months
  Change of skeletal muscle index (SMI) between both groups.

SECONDARY OUTCOMES:
Number of patients who improved sarcopenia in encourage using pedometer group and discourage using pedometer group. | 6 months
  Number of sarcopenic patient improvement in both groups
Mortality rate in encourage using pedometer group and discourage using pedometer group. | 12 months
  Mortality rate in both groups
The hospital admission | 12 months
  hospital admission in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Witchuta Niamsanit, Gastroenterologist, Principal Investigator — Siriraj Hospital
Locations (1):
- Witchuta Niamsanit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Montano-Loza AJ, Meza-Junco J, Prado CM, Lieffers JR, Baracos VE, Bain VG, Sawyer MB. Muscle wasting is associated with mortality in patients with cirrhosis. Clin Gastroenterol Hepatol. 2012 Feb;10(2):166-73, 173.e1. doi: 10.1016/j.cgh.2011.08.028. Epub 2011 Sep 3. PMID 21893129
- [Background] Kalafateli M, Konstantakis C, Thomopoulos K, Triantos C. Impact of muscle wasting on survival in patients with liver cirrhosis. World J Gastroenterol. 2015 Jun 28;21(24):7357-61. doi: 10.3748/wjg.v21.i24.7357. PMID 26139982
- [Background] Volpi E, Nazemi R, Fujita S. Muscle tissue changes with aging. Curr Opin Clin Nutr Metab Care. 2004 Jul;7(4):405-10. doi: 10.1097/01.mco.0000134362.76653.b2. PMID 15192443
- [Background] Hiraoka A, Michitaka K, Kiguchi D, Izumoto H, Ueki H, Kaneto M, Kitahata S, Aibiki T, Okudaira T, Tomida H, Miyamoto Y, Yamago H, Suga Y, Iwasaki R, Mori K, Miyata H, Tsubouchi E, Kishida M, Ninomiya T, Kohgami S, Hirooka M, Tokumoto Y, Abe M, Matsuura B, Hiasa Y. Efficacy of branched-chain amino acid supplementation and walking exercise for preventing sarcopenia in patients with liver cirrhosis. Eur J Gastroenterol Hepatol. 2017 Dec;29(12):1416-1423. doi: 10.1097/MEG.0000000000000986. PMID 29016470
- [Background] Ismaiel A, Bucsa C, Farcas A, Leucuta DC, Popa SL, Dumitrascu DL. Effects of Branched-Chain Amino Acids on Parameters Evaluating Sarcopenia in Liver Cirrhosis: Systematic Review and Meta-Analysis. Front Nutr. 2022 Jan 27;9:749969. doi: 10.3389/fnut.2022.749969. eCollection 2022. PMID 35155535
- [Background] Konstantis G, Pourzitaki C, Chourdakis M, Kitsikidou E, Germanidis G. Efficacy of branched chain amino acids supplementation in liver cirrhosis: A systematic review and meta-analysis. Clin Nutr. 2022 Jun;41(6):1171-1190. doi: 10.1016/j.clnu.2022.03.027. Epub 2022 Apr 1. PMID 35500317
- [Background] Harper AE, Miller RH, Block KP. Branched-chain amino acid metabolism. Annu Rev Nutr. 1984;4:409-54. doi: 10.1146/annurev.nu.04.070184.002205. No abstract available. PMID 6380539
- [Background] Roman E, Torrades MT, Nadal MJ, Cardenas G, Nieto JC, Vidal S, Bascunana H, Juarez C, Guarner C, Cordoba J, Soriano G. Randomized pilot study: effects of an exercise programme and leucine supplementation in patients with cirrhosis. Dig Dis Sci. 2014 Aug;59(8):1966-75. doi: 10.1007/s10620-014-3086-6. Epub 2014 Mar 6. PMID 24599772
- [Background] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811
- [Background] Dunn MA, Kappus MR, Bloomer PM, Duarte-Rojo A, Josbeno DA, Jakicic JM. Wearables, Physical Activity, and Exercise Testing in Liver Disease. Semin Liver Dis. 2021 May;41(2):128-135. doi: 10.1055/s-0040-1716564. Epub 2021 Jan 14. PMID 33788206
- [Background] Dunn MA, Josbeno DA, Schmotzer AR, Tevar AD, DiMartini AF, Landsittel DP, Delitto A. The gap between clinically assessed physical performance and objective physical activity in liver transplant candidates. Liver Transpl. 2016 Oct;22(10):1324-32. doi: 10.1002/lt.24506. PMID 27348200
- [Background] Ross R, Blair SN, Arena R, Church TS, Despres JP, Franklin BA, Haskell WL, Kaminsky LA, Levine BD, Lavie CJ, Myers J, Niebauer J, Sallis R, Sawada SS, Sui X, Wisloff U; American Heart Association Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Cardiovascular and Stroke Nursing; Council on Functional Genomics and Translational Biology; Stroke Council. Importance of Assessing Cardiorespiratory Fitness in Clinical Practice: A Case for Fitness as a Clinical Vital Sign: A Scientific Statement From the American Heart Association. Circulation. 2016 Dec 13;134(24):e653-e699. doi: 10.1161/CIR.0000000000000461. Epub 2016 Nov 21. PMID 27881567
- [Background] Singh Tejavath A, Mathur A, Nathiya D, Singh P, Raj P, Suman S, Mundada PR, Atif S, Rai RR, Tomar BS. Impact of Branched Chain Amino Acid on Muscle Mass, Muscle Strength, Physical Performance, Combined Survival, and Maintenance of Liver Function Changes in Laboratory and Prognostic Markers on Sarcopenic Patients With Liver Cirrhosis (BCAAS Study): A Randomized Clinical Trial. Front Nutr. 2021 Sep 22;8:715795. doi: 10.3389/fnut.2021.715795. eCollection 2021. PMID 34631765
- [Background] Aamann L, Dam G, Borre M, Drljevic-Nielsen A, Overgaard K, Andersen H, Vilstrup H, Aagaard NK. Resistance Training Increases Muscle Strength and Muscle Size in Patients With Liver Cirrhosis. Clin Gastroenterol Hepatol. 2020 May;18(5):1179-1187.e6. doi: 10.1016/j.cgh.2019.07.058. Epub 2019 Aug 5. PMID 31394282
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Degroote L, Hamerlinck G, Poels K, Maher C, Crombez G, De Bourdeaudhuij I, Vandendriessche A, Curtis RG, DeSmet A. Low-Cost Consumer-Based Trackers to Measure Physical Activity and Sleep Duration Among Adults in Free-Living Conditions: Validation Study. JMIR Mhealth Uhealth. 2020 May 19;8(5):e16674. doi: 10.2196/16674. PMID 32282332
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Result] Duarte-Rojo A, Ruiz-Margain A, Montano-Loza AJ, Macias-Rodriguez RU, Ferrando A, Kim WR. Exercise and physical activity for patients with end-stage liver disease: Improving functional status and sarcopenia while on the transplant waiting list. Liver Transpl. 2018 Jan;24(1):122-139. doi: 10.1002/lt.24958. PMID 29024353
- [Result] Lin FP, Bloomer PM, Grubbs RK, Rockette-Wagner B, Tevar AD, Dunn MA, Duarte-Rojo A. Low Daily Step Count Is Associated With a High Risk of Hospital Admission and Death in Community-Dwelling Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1813-1820.e2. doi: 10.1016/j.cgh.2022.03.012. Epub 2022 Mar 21. PMID 35331941
- [Result] Pino-Ortega J, Gomez-Carmona CD, Rico-Gonzalez M. Accuracy of Xiaomi Mi Band 2.0, 3.0 and 4.0 to measure step count and distance for physical activity and healthcare in adults over 65 years. Gait Posture. 2021 Jun;87:6-10. doi: 10.1016/j.gaitpost.2021.04.015. Epub 2021 Apr 15. PMID 33866152
- [Result] Cichoz-Lach H, Michalak A. A Comprehensive Review of Bioelectrical Impedance Analysis and Other Methods in the Assessment of Nutritional Status in Patients with Liver Cirrhosis. Gastroenterol Res Pract. 2017;2017:6765856. doi: 10.1155/2017/6765856. Epub 2017 Aug 13. PMID 28894465